CLINICAL TRIAL: NCT00646464
Title: New Computerized Continuous Performance Test (CPT) for Diagnosing Pediatric Attention Deficit/Hyperactivity Disorder (ADHD)
Brief Title: New Continuous Performance Tests (CPT) for the Diagnosis of Pediatric Attention Deficit/Hyperactivity Disorder (ADHD)
Acronym: CPT
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0052-08-HMO-CTIL
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2009-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: CPT; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 2: Children 6-12 years old diagnosed as not suffering from ADHD
- 1: children 6-12 diagnosed as ADHD

SUMMARY:
Computerized continuous performance tests (CPT) considered the "gold standard" for diagnosis of Attention Deficit/Hyperactivity Disorder (ADHD.

This type of tests are based mainly on visual performance. The available tests suffer from high false negative errors. This raises questions regarding their ability to correctly diagnose ADHD.

With the expanding knowledge regarding the neurobiological basis in ADHD we have learned that attention is not a general property of the whole brain, but involves several coordinated networks. This knowledge promoted us to the stage in which we can recognize different types of attention domains.

Our diagnosis test can separate between the different attention abilities and provide specific diagnosis. Our program is individually fits for the specific child difficulties and covers a wider range of needs. So, it can be helpful to a larger variety of children with different needs.

DETAILED DESCRIPTION:
Computerized continuous performance tests (CPT) considered the "gold standard" for diagnosis of Attention Deficit/Hyperactivity Disorder (ADHD) and are widely used.

This type of tests measures the number of correctly detected stimuli as well as response time. The diagnosis in this tests based mainly on visual performance. The available tests in the market suffer from high false negative errors. In some subgroups of children the error can be false positive. All this raises questions regarding their ability to correctly diagnose ADHD. There are also doubts regarding the validity of these tests. From the medical literature and from our own experience it seems that with the current tests as much as third of the children who fulfill DSM criteria for ADHD can escape detection.

With the expanding knowledge regarding the neurobiological basis in ADHD we have learned that attention is not a general property of the whole brain, but involves several coordinated networks. These networks must be orchestrated in order to perform normally in three main domains of attention = alertness, orientation and executive function. This raised the need for a better, more accurate and valid computerized test.

This knowledge promoted us to the stage in which we can recognize different types of attention domains. We can separate between - visual attention, auditory attention, spatial attention, integrated attention, sustained attention, covert and overt attention, working memory, the ability to integrate and disintegrate attention, attention span, focusing, impulsivity and response time. Different people have different "subtypes" of ADHD. The individual separation and ability to focus on specific difficulties influence diagnosis process and treatment methods.

Our diagnosis test can separate between the different attention abilities and provide the parents with specific diagnosis of their child and in this way direct them to the appropriate diagnosis and treatment. Moreover, we expect its falls negative and positive errors to be negligible.

The next phase - involves training and exercise. It is proved that training can improve attention.

We have also developed a computerized training program for children. This program is based on the same platform as the diagnosis test and can recommend on training in the individual difficulties of the specific child.

Other programs are already distributed in the market for the same propose. The other programs focus on improving a general specific skill and ignore (or can not focus) on the specific need of the individual. They can try to improve working memory which is only one aspect in attention domain. Or, based on improving visual-motor skill, which is a skill that can be improved in regular computer games and again focus on a specific short range difficulty. In many children ADHD symptoms and signs are due to other sources. For them improving working memory or visual-motor skills will not change their every day performance.

Our program is better since it is individually fits for the specific child difficulties and covers a wider range of needs. So, it can be helpful to a larger variety of children with different needs.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ADHD by the "gold standard" method

Exclusion Criteria:

* Chronic use of medications, Psychiatric disorder, Abnormal cognitive function

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 6-12 year old children suspected as ADHD otherwise healthy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
accurate diagnosis of ADHD | one year

SECONDARY OUTCOMES:
validation | one year

CONTACTS AND LOCATIONS:
Overall Officials: Itai Berger, MD, Principal Investigator — Hadassah Medical Organization
Locations (2):
- Israel (2):
  - Neuro-Pediatric Unit, Hadassah-Hebrew University Medical Center Mount Scopus, Jerusalem
  - Neuro-Pediatric Unit, Hadassah-Hebrew University Medical Center, Jerusalem

REFERENCES:
- [Background] Rueda MR, Rothbart MK, McCandliss BD, Saccomanno L, Posner MI. Training, maturation, and genetic influences on the development of executive attention. Proc Natl Acad Sci U S A. 2005 Oct 11;102(41):14931-6. doi: 10.1073/pnas.0506897102. Epub 2005 Sep 28. PMID 16192352
- [Background] Lee HJ, Cho S, Shin MS. Supporting diagnosis of attention-deficit hyperactive disorder with novelty detection. Artif Intell Med. 2008 Mar;42(3):199-212. doi: 10.1016/j.artmed.2007.11.001. Epub 2008 Jan 9. PMID 18187311